CLINICAL TRIAL: NCT05723510
Title: An Open-label, Randomized, Crossover Study to Evaluate the Pharmacokinetic and Pharmacodynamic Interaction Between Tegoprazan and Novel Oral Anticoagulants (NOACs) After Multiple Oral Dosing in Healthy Volunteers
Brief Title: PK and PD Interaction Between Tegoprazan and NOACs After Multiple Oral Dosing in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: HK inno.N Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IN_APA_121
Record Dates: First submitted 2023-02-02; First posted 2023-02-10 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Healthy
MeSH Terms: interventions — tegoprazan; edoxaban; apixaban; Rivaroxaban

STUDY DESIGN:
Intervention Model Description: two-arm, two-period crossover
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Edoxaban 60mg (Experimental): Multiple dosing of edoxaban alone once daily for 5 days
  Interventions: Drug: Edoxaban 60mg
- Edoxaban 60mg + Tegoprazan 50mg (Experimental): Multiple dosing of edoxaban once daily in combination with tegoprazan once daily for 5 days
  Interventions: Drug: Tegoprazan 50mg; Drug: Edoxaban 60mg
- Apixaban 5mg (Experimental): Multiple dosing of apixaban alone twice daily for 5 days
  Interventions: Drug: Apixaban 5mg
- Apixaban 5mg + Tegoprazan 50mg (Experimental): Multiple dosing of apixaban twice daily in combination with tegoprazan once daily for 5 days
  Interventions: Drug: Tegoprazan 50mg; Drug: Apixaban 5mg
- Rivaroxaban 20mg (Experimental): Multiple dosing of rivaroxaban alone once daily for 5 days
  Interventions: Drug: Rivaroxaban 20mg
- Rivaroxaban 20mg + Tegoprazan 50mg (Experimental): Multiple dosing of rivaroxaban once daily in combination with tegoprazan once daily for 5 days
  Interventions: Drug: Tegoprazan 50mg; Drug: Rivaroxaban 20mg

INTERVENTIONS:
Drug: Tegoprazan 50mg — Oral administration of one tablet of tegoprazan 50 mg once daily
  Other Names: K-CAB Tab. 50 mg
  Arms: Apixaban 5mg + Tegoprazan 50mg; Edoxaban 60mg + Tegoprazan 50mg; Rivaroxaban 20mg + Tegoprazan 50mg
Drug: Edoxaban 60mg — Oral administration of one tablet of edoxaban 60 mg once daily
  Other Names: Lixiana Tab. 60mg
  Arms: Edoxaban 60mg; Edoxaban 60mg + Tegoprazan 50mg
Drug: Apixaban 5mg — Oral administration of one tablet of apixaban 5 mg twice daily
  Other Names: Eliquis Tab. 5 mg
  Arms: Apixaban 5mg; Apixaban 5mg + Tegoprazan 50mg
Drug: Rivaroxaban 20mg — Oral administration of one tablet of rivaroxaban 20 mg once daily
  Other Names: Xarelto Tab. 20 mg
  Arms: Rivaroxaban 20mg; Rivaroxaban 20mg + Tegoprazan 50mg

SUMMARY:
This study aims to evaluate the effects of combination therapy of tegoprazan and novel oral anticoagulants (NOACs) on the pharmacokinetic and pharmacodynamic properties of NOACs in healthy adults.

DETAILED DESCRIPTION:
A randomized, open-label, multiple-dose, two-arm, two-period crossover study

[Cohort 1] To evaluate the effects of combination therapy of tegoprazan and edoxaban on the pharmacokinetic and pharmacodynamic properties of edoxaban in healthy adults.

[Cohort 2] To evaluate the effects of combination therapy of tegoprazan and apixaban on the pharmacokinetic and pharmacodynamic properties of apixaban in healthy adults.

[Cohort 3] To evaluate the effects of combination therapy of tegoprazan and rivaroxaban on the pharmacokinetic and pharmacodynamic properties of rivaroxaban in healthy adults.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adults aged ≥ 19 years to < 55 years at the time of screening
2. Those with body weight ≥ 45 kg (but ≥ 60 kg for cohort 1 and cohort 2) and body mass index (BMI) in the range of 19.0 kg/m2 to 27.0 kg/m2 at the time of screening

   ☞ BMI = weight (kg) / height (m)2
3. Those who have neither congenital/chronic disease (within recent 3 years) nor pathological symptoms/findings as a result of medical examination
4. Those determined to be eligible for this study based on the findings of screening such as clinical laboratory tests (hematological test, blood chemistry test, blood coagulation test, urinalysis, test for viruses/bacteria, etc.), vital signs, and electrocardiogram (ECG) which are performed by the investigator according to the properties of medicines
5. Those who are fully informed of study purpose, procedures, etc., voluntarily decide to participate in this study, and sign an informed consent form (ICF) approved by the Institutional Review Board (IRB) of Jeonbuk National University Hospital, prior to participation in the study
6. Those with a capability/willingness to participate throughout the study

Exclusion Criteria:

1. Medical history of clinically significant blood, renal, endocrine, respiratory, gastrointestinal (peptic ulcer, etc.), urinary, cardiovascular, hepatic, psychiatric, neurological or immune disease (but except for history of simple dental treatment such as tartar, impacted teeth, and third molar teeth) or evidence thereof
2. Previous history of gastrointestinal disease (except for esophageal disease such as esophageal achalasia or esophageal stricture, inflammatory bowel disease (Crohn's disease, ulcerative colitis)) or surgery (not including simple appendectomy, hernia surgery, tooth extraction, etc.) which may affect drug absorption
3. Following findings of clinical laboratory tests:

   ☞ ALT or AST value > twice the upper limit of normal (ULN)
4. History of periodic alcohol consumption exceeding 210 g/week within 6 months prior to screening (beer (5%) 1 glass (250 mL) = 10 g, soju (20%) 1 glass (50 mL) = 8 g, wine (12%) 1 glass (125 mL) = 12 g)
5. Administration of another investigational product within 6 months prior to the first dose of the investigational product
6. History of serious alcohol or drug misuse and abuse within 1 year prior to screening
7. Administration of drugs known to markedly induce or inhibit drug metabolizing enzymes within 30 days prior to the first dose of the investigational product
8. History of smoked cigarettes ≥ 20 cigarettes/day within 6 months prior to screening
9. Administration of a prescription or non-prescription drug within 10 days prior to the first dose of the investigational product
10. Whole blood donation within 2 months prior to the first dose of the investigational product or apheresis donation within 1 month prior to the first dose of the investigational product
11. Those who may be put at an increased risk due to the adminisration of the investigational product and study participation or have a severe acute/chronic medical or mental condition which may interfere with the interpretation of study results
12. Patients with hypersensitivity to tegoprazan, edoxaban, apixaban, rivaroxaban, etc. (e.g., asthma, acute rhinitis, nasal polyp, angioedema, urticaria, allergic reactions, etc.)
13. Patients with a clinically significant bleeding
14. Patients with hemostatic disorder and hepatic disease related to a clinically significant risk of bleeding
15. Severe hepatic impairment
16. Renal impairment (eGFR <60 ml/min/1.73m2)
17. Hereditary problems such as galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption
18. Pregnant/breast-feeding women
19. Those who cannot use medically acceptable contraceptive methods throughout the study

    ▶ Medically acceptable contraceptive methods
    * Use of intrauterine device (IUD) showing a demonstrated pregnancy failure rate
    * Combined use of barrier contraceptive method (for male or female) and spermicide
    * Use of vasectomy, tubectomy/tubal ligation, or hysterectomy
20. Those who are not eligible for the study in the judgment of the investigator

Ages: 19 Years to 54 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 87 (Actual)
Dates: Start 2023-03-06 (Actual); Primary Completion 2023-07-17 (Actual); Study Completion 2023-07-24 (Actual)

PRIMARY OUTCOMES:
AUCτ and Css,max of edoxaban | Pre-dose(0 hour) on 1D, 3D, and 4D for each period; pre-dose(0 hour) up to 48 hours after treatment on 5D for each period
  Area under the plasma concentration-time curve during a steady-state dosing interval (τ) and maximum plasma concentration at steady state of edoxaban
AUCτ and Css,max of apixaban | Pre-dose (0 hour) in the morning on 1D and in the morning and afternoon on 4D for each period; pre-dose(0 hour) in the morning up to 48 hours after treatment on 5D for each period
  Area under the plasma concentration-time curve during a steady-state dosing interval (τ) and maximum plasma concentration at steady state of apixaban
AUCτ and Css,max of rivaroxaban | Pre-dose (0 hour) on 1D, 3D, and 4D for each period; pre-dose(0 hour) up to 48 hours after treatment on 5D for each period
  Area under the plasma concentration-time curve during a steady-state dosing interval (τ) and maximum plasma concentration at steady state of rivaroxaban
AUECτ and Emax of Anti-Factor Xa activity, PT, aPTT, and Prothrombin (INR) | Pre-dose (0 hour) up to 24 hours after treatment on 5D for each period
  Area under the effect-time curve over the dosing interval (τ) at steady state and maximum effect of Anti-Factor Xa activity, PT, aPTT, and Prothrombin (INR)

CONTACTS AND LOCATIONS:
Overall Officials: Min-Gul Kim, Principal Investigator — Clinical Pharmacology Center, Jeonbuk National University Hospital
Locations (1):
- Jeonbuk National University Hospital, Jeonju, South Korea